CLINICAL TRIAL: NCT01401348
Title: The Stanford HIV Aging Cohort (SHAC)
Brief Title: Stanford Universities: The Stanford HIV Aging Cohort
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Philip Grant, Principal Investigator, Stanford University
Other Study IDs: SU-12142010-7318
Record Dates: First submitted 2011-07-19; First posted 2011-07-25 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC's
Oversight: Data Monitoring Committee: No

SUMMARY:
A research study to evaluate the effect of aging and HIV on neurocognitive dysfunction (declining ability to process information), physical frailty and heart disease. HIV-infected participants whose virus is controlled on antiretroviral medications will be studied to determine the rates and risk factors of developing these conditions.

DETAILED DESCRIPTION:
With advances in antiretroviral therapy, the life expectancy of HIV-infected individuals continues to improve with older individuals representing a rapidly growing proportion of those infected. However, despite improved life expectancy, substantial residual morbidity remains in treated HIV including increased rates of neurocognitive dysfunction, frailty, and cardiovascular disease. As these conditions also increase with normal aging, HIV is often thought to be a risk factor for "early" or "accelerated" aging. Prior studies have generally focused on HIV-specific factors and risk for neurocognitive dysfunction, frailty, and cardiovascular disease, while few have examined extensively risk factors found to be significant for these conditions in the general population.

The investigators hypothesize that the effects of age and HIV will be synergistic on the rates of non-AIDS morbidity. While the correlates and risk factors for non-AIDS morbidity in younger individuals may largely be related to HIV, in older individuals with sustained virologic control, traditional risk factors for neurocognitive disease, frailty, and cardiovascular disease will contribute more significantly to disease than HIV-specific risk factors. Our primary objectives are to:

1. Define the prevalence and incidence of neurocognitive dysfunction, frailty, and cardiovascular disease in a well-defined cohort of aging virologically suppressed HIV-infected individuals.
2. Identify correlates and risk factors for prevalent and incident neurocognitive dysfunction, frailty, and cardiovascular disease.
3. Compare and contrast the identified correlates and risk factors for the co-morbidities of interest in older (>50 years old) and younger HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an HIV RNA level below the limit of quantification (e.g., <75 copies, <50 copies, or <48 copies/mL, depending on the assay used) for at least 6 months excluding "blips" (e.g., a single measurement between 48-200 copies/mL preceded and followed by measurements below the limit of quantification) while on antiretroviral therapy.

Exclusion Criteria:

1. Completed treatment for any acute systemic infection (other than HIV-1) less than four weeks before study entry.
2. Any active brain infection (except for HIV-1), brain neoplasm, or space-occupying brain lesion.
3. Receipt of immunomodulating medication (e.g., corticosteroids, immunoglobulin, etc.) within four weeks of study entry.
4. Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound the analysis of the neuropsychological test results.
5. Active drug or alcohol abuse that, in the investigator's opinion, could prevent compliance with study procedures or confound the analysis of study endpoints.
6. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 HIV-infected participants whose virus is controlled on antiretroviral medications from the Stanford Positive Care Clinic. Five (150) patients over 50 years old and five (150) patients less than 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
neurocognitive testing | 1 year
  Controlled oral word association test-FAS, Paced auditory serial addition task, trail making a and b, REY auditory verbal learning test, grooved peg board, timed gait

SECONDARY OUTCOMES:
cardiovascular testing | 1 yr
  ankle-brachial index

CONTACTS AND LOCATIONS:
Overall Officials: Philip Grant, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States